CLINICAL TRIAL: NCT04648488
Title: Early Mobilisation After Surgery in Patients With Elbow Fracture-dislocation - a Randomised Clinical Trial
Brief Title: Early Mobilisation After Surgery in Patients With Elbow Fracture-dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Östergötland (Other)
Collaborators: Kalmar County Council (Unknown); Jönköping county council (Unknown)
Responsible Party: Principal Investigator, Teresa Holmgren, PhD Registered physiotherapist, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202004709
Record Dates: First submitted 2020-10-26; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Early Mobilization; Elbow Stiffnes; Elbow Fracture
Keywords: Upper extremity function; Elbow stiffnes; Early mobilization
MeSH Terms: conditions — Elbow Fractures

STUDY DESIGN:
Intervention Model Description: Randomised Clinical trail
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early mobilisation (Experimental): Patients will start unloaded exercise treatment 3 days after surgery. They will remove the plaster 5 times every day to perform range of motion exercises.
  Interventions: Other: Experimental early mobilisation
- Standard treatment (Active Comparator): Patients will have a plaster 3 weeks after surgery and after that start with exercise treatment.
  Interventions: Other: Aktive comparator standrad treatmnet

INTERVENTIONS:
Other: Experimental early mobilisation — early activ assisted exercises treatment
  Arms: Early mobilisation
Other: Aktive comparator standrad treatmnet — standard treatment with a plaster 3 weeks and then active assisted exercises
  Arms: Standard treatment

SUMMARY:
The purpose with the study is to evalute if early mobilsation after surgery in patients vid elbow frakture-dislocation may lead to better armfunction and reduce common complications as stiffnes in the elbow. After surgery patients will be randomised to either early mobilisation (exercise treatment 3 Days after surgery) or ordinary treatment (plaster and exercise treatment 3 weeks after surgery).

DETAILED DESCRIPTION:
In patients with elbow fracture in combinations with dislocation, surgery is often indicated. After surgery the ordinary standard praxis treatment is immobilisation in a plaster for 3 weeks. One common complication is "stiff elbow". Stiffness in the elbow may be due to "heterotopic ossification" which is the abnormal growth of bone in the non-skeletal tissues including muscles or tendons. There is a prospective study that have reported positive results with early mobilisation starting two days after surgery in these patients. However, randomised clinical trials are missing. Therefore our aim was to investigate if early mobilisation may increase elbow function (increased range of motion and decreased pain) and also reduce comlications as stiff elbow compared to ordinary treatment in these patients.

All patients operated with elbow fracture-dislocation at the University hospital in Linköping were asked if the wanted to participate in the study. They had thourough written and oral information about the study. If they agree to participate written informed consent was collected. After surgery patients were randomised to either early mobilisation or to ordinary treatment (standard praxis).

At baseline before surgery or directly after patients filled in some background vatiables such as gender, age social status medical treatment etc They also filled in some self-adminstrated outcome measure in purpuse to evalute upper extremity function and activity and health related quality of Life.

Follow ups with X ray and upper extremity function and activity were at 3 weeks 3 and 12 months with an independent observer.

In beteween these follow ups patient followed the treatment regime (ordinary or early exrecise treatment) and had support from a physiotherapist.

ELIGIBILITY:
Inclusion Criteria: Patients over 18 years with elbow fracture-dislocation being operated on.

-

Exclusion Criteria:

* ongoing cancer and earlier radiation therapy in the study arm
* neurological disease
* cervcialgia or disc herniation in the neck
* associated nerv or blodvessel injury
* dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Oxford elbow score (OES 0-48 Points) | 12 month follow up
  Evaluating pain, elbowfunction and psychological status

SECONDARY OUTCOMES:
upper extremity activity scale (0-8) | 12 month follow up
  Activity level Before and after injury
Range of motion | 12 month follow up
  elbow range of motion measured with goniometer
Heterotopic ossification | 3 month follow up
  Number of patients with heterotopic ossification verfified by X ray
Re-operation | in between 3 and 12 month follow up
  Number of patients with stiff elbow who need re-operation
Patient Global impression of change | at three and 12 months
  Patient satisfaction

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-05-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT04648488/Prot_000.pdf